CLINICAL TRIAL: NCT05680337
Title: Transcutaneous Electrical Auricular Vagus Stimulation and Heart Rate Variability
Brief Title: Auricular Vagus Stimulation and Heart Rate Variability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Collaborators: State Budget Public Health Institution Scientific Research Institute - Ochapovsky Regional Clinical Hospital (Other Government); Astrakhan Federal Centre For Cardiac Surgery (Other)
Responsible Party: Principal Investigator, Vladimir A Shvartz, MD, MD, DM, Professor, Bakulev Scientific Center of Cardiovascular Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: #6
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Vagus Nerve Stimulation; Heart Rate Variability
Keywords: auricular stimulation; auricular vagus nerve stimulation; heart rate; transcutaneous vagus nerve stimulation (TENS); vagus nerve stimulation (VNS); heart rate variability; power of high-frequency oscillations (HF); power of low-frequency oscillations (LF); power of very low frequency oscillations (VLF); power of ultra-low frequency oscillations (ULF); LF/HF; index centralization (IC); index of vegetative balance (IVB)
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of active stimulation vs. sham stimulation
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS (Active Comparator): Active will be performed with using a TENS device with an ear clip attached to the tragus of the left ear (which is innervated by auricular branch of the vagus nerve) at 20 Hz, 200 μs at a current just below discomfort threshold.
  Interventions: Device: TENS
- Sham TENS (Sham Comparator): Sham will be performed with using a TENS device with an ear clip attached to the left earlobe (which is devoid of vegas innervation) at 20 Hz, 200 μs at a current just below discomfort threshold.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — TENS stimulation will occur within 10 minutes. HRV parameters will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.

SUMMARY:
Transcutaneous electrical stimulation of the auricular vagus nerve (TENS) is a promising method of neuromodulation of the autonomic nervous system in patients with various pathologies. The use of this method requires the determination of a reliable biomarker of successful activation of the vagus nerve using TENS. Currently, most studies focus on the assessment of heart rate variability (HRV) as a marker of the functioning of the autonomic nervous system.

Despite the physiological justification of HRV as a biomarker for TENS, the data on the effects of TENS on HRV are ambiguous. In some studies, a significant decrease in the ratio of spectral characteristics (LF/HF) in active TENS was found in comparison with fictitious stimulation (sham), which indicated an increase in the parasympathetic component of HRV. However, other studies have not revealed an increase in HRV.

DETAILED DESCRIPTION:
Transcutaneous vagus nerve stimulation (TENS) involves the stimulation of the left and/or right auricular branch of the vagus nerve in the area of the cymba concha with low-frequency electrical impulses. The auricular branch of the vagus nerve runs superficially, which makes it a favorable target for non-invasive stimulation techniques to modulate vagal activity. It gained popularity due to minimal side effects and low cost.

This method is a new, cost-effective alternative to invasive cervical vagus nerve stimulation (iVNs), which is an FDA-approved treatment of depression resistant to the treatment, epilepsy and other pathologies.

The use of TENS has shown similar positive results as iVNs, for example, in reducing symptoms in patients with depression and changing the early visual processing of negative emotional stimuli in adolescent depression. Similarly, positive effects of TENS have also been found in chronic pain and epilepsy. These similarities in effects can be explained by the similarity of brain network activation achieved by iVNs and TENS.

The lack of similarity between behavioral studies and numerous theories of physiological processes in TENS make it necessary to determine a reliable biomarker of successful activation of the vagus nerve using TENS. Although many potential biomarkers have been proposed, most studies have focused on HRV.

Despite the physiological justification of HRV as a biomarker for TENS, the data on the effects of TENS on HRV are ambiguous. In some studies, a significant decrease in the ratio of spectral characteristics (LF/HF) in active TENS compared to fictitious stimulation (sham) was found, indicating an increase in the parasympathetic component of HRV.

However, other studies have not revealed an increase in HRV. Large methodological differences between studies, such as different stimulation devices, sides and places of stimulation, experimental schemes, reported HRV parameters and stimulation protocols, reduce comparability between studies.

One of the most striking examples is the use of various control conditions. While in most studies active TENS are compared with imitation of the earlobe as an independent variable, as recommended, in some studies active stimulation of the tragus was compared with a control state without stimulation or with a fictitious state without stimulation when the electrode is placed on the ear, but no electric current is applied.

The development of international agreed consensus guidelines on TENS research reporting should address these issues. Although TENS represents a potential treatment option for many disorders and it is an interesting tool for experimental research, it needs to be studied in an objective and reliable way before its true place as a neuro-immunomodulatory intervention can be determined.

The investigators plan to conduct a study on the assessment of TENS on the dynamics of HRV parameters with reporting according to the international consensus document https://www.frontiersin.org/articles/10.3389/fnhum.2020.568051/full#B235

ELIGIBILITY:
Inclusion Criteria:

* Sinus rhythm at the time of registration

Exclusion Criteria:

* Frequent ventricular / supraventricular extrasystole, 2d/3d degree AV Block
* Taking glucocorticosteroids in the last 1 month
* Taking any antiarrhythmics, except beta blockers
* Severe chronic renal or liver pathology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Dynamics of LF/HF | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of LF /HF relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation

SECONDARY OUTCOMES:
HR dynamics | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the HR level relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation
Dynamics of SDNN | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of SDNN relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation
Dynamics of IVB | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of IVB relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation
Dynamics of IC1 | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of IC1 relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation. IC1 (Index Centralization) = (HF+LF)/VLF
Dynamics of IC2 | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of IC2 relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation. IC2 (Index Centralization) = (VHF+LF)/LF
Dynamics of HF% | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of HF% relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation
Dynamics of LF% | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of LF% relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation
HF dynamics | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the HF level relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation
Dynamics of LF | This parameter will be evaluated before stimulation initially at rest, in the first 5 minutes of stimulation, in the second 5 minutes of stimulation and after the end of stimulation.
  Changes in the level of LF relative to the initial and after the end of stimulation in the groups of active and fictitious stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Shvartz, Principal Investigator — Bakoulev Scientific Center for Cardiovascular Surgery
Locations (3):
- Russia (3):
  - Federal Center for Cardiovascular Surgery (Astrakhan), Astrakhan
  - State Budget Public Health Institution Scientific Research Institute - Ochapovsky Regional Clinical Hospital, Krasnodar
  - Bakulev National Medical Research Center for Cardiovascular Surgery, Moscow

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed during the current study are publicly available. The data is available in the general repository "Open Science Framework" at the link
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2023
Access Criteria: open access
URL: https://doi.org/10.17605/OSF.IO/STU62

REFERENCES:
- [Result] Shvartz, V.; Sizhazhev, E.; Sokolskaya, M.; Koroleva, S.; Enginoev, S.; Kruchinova, S.; Shvartz, E.; Golukhova, E. The Effect of Short-Term Transcutaneous Electrical Stimulation of Auricular Vagus Nerve on Parameters of Heart Rate Variability. Data 2023, 8, 87. https://doi.org/10.3390/data8050087
- [Result] Shvartz V.A., Sizhazhev E.M. Percutaneous stimulation of the auricular branch of the vagus: the potential of the method of treatment of different cardiovascular diseases. Clinical Physiology of Circulation. 2023; 20 (1): 5-15 (in Russ.). DOI: 10.24022/1814-6910-2023-20-1-5-15
- See also: International Consensus Based Review and Recommendations for Minimum Reporting Standards in Research on Transcutaneous Vagus Nerve Stimulation (Version 2020) — https://doi.org/10.3389/fnhum.2020.568051
- See also: Toward Diverse or Standardized: A Systematic Review Identifying Transcutaneous Stimulation of Auricular Branch of the Vagus Nerve in Nomenclature — https://doi.org/10.1111/ner.13346
- See also: Does transcutaneous auricular vagus nerve stimulation affect vagally mediated heart rate variability? A living and interactive Bayesian meta-analysis — https://www.biorxiv.org/content/10.1101/2021.01.18.426704v1.full